CLINICAL TRIAL: NCT06808516
Title: The OxyPLEASURE Study - Effects of Intranasal Oxytocin on Sexual Well-Being in Patients With Arginine Vasopressin Deficiency (Central Diabetes Insipidus) and Healthy Controls - a Double-blind Randomized Placebo-controlled Crossover Trial
Brief Title: Effects of Intranasal Oxytocin on Sexual Well-Being in Patients With Arginine Vasopressin Deficiency and Healthy Controls
Acronym: OxyPLEASURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02116; kt24ChristCrain4
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Arginine Vasopressin Deficiency; Central Diabetes Insipidus; Oxytocin Deficiency
Keywords: Nasal oxytocin; Sexual Well-Being
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: This randomized, placebo-controlled trial with a double-blind, cross-over design examines patients with AVP-D compared to healthy controls.
  * Part A investigates the acute effects of intranasal OXT on sexual well-being and intimacy during intercourse over a seven-day treatment period in couples where one partner has AVP-D, compared to healthy couples. Using a cross-over design with a three-week washout aligned to the female participant's menstrual cycle, only couples in stable relationships are eligible. Participants complete self-evaluations at baseline and after each treatment period.
  * Part B, conducted in a clinical setting, includes single participants and those in relationships. It assesses subjective sexual arousal, fear perception, empathy, and physical and hormonal responses to visual stimuli following intranasal OXT or placebo. Randomized participants receive a single application of OXT or placebo, with a 72-hour or three-week washout depending on study participation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The OXT and placebo nasal spray will be identical in volume, labelling and container systems, so that they cannot be differentiated from one another. The placebo will contain no OXT but 0.9% normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oxy part A: 7 Day treatment (Experimental): Syntocinon, 24 IU, administered over a 7 day period
  Interventions: Drug: Oxytocin nasal spray
- Placebo part A: 7 Day treatment (Placebo Comparator): 0.9% sodium chloride, administered over a 7 day period
  Interventions: Drug: Placebo
- Oxy part B: single application (Experimental): Syntocinon, 24 IU, administered once
  Interventions: Drug: Oxytocin nasal spray
- Placebo Oxy part B: single application (Placebo Comparator): 0.9% sodium chloride, administered once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — 24 IU
  Other Names: Syntocinon
  Arms: Oxy part A: 7 Day treatment; Oxy part B: single application
Drug: Placebo — 0.9% NaCl
  Arms: Placebo Oxy part B: single application; Placebo part A: 7 Day treatment

SUMMARY:
The study aims to investigate whether intranasal oxytocin (OXT) improves sexual well-being in patients with Arginine Vasopressin Deficiency (AVP-D). The trial consists of two parts: Part A assesses the effect of OXT on sexual well-being and intimacy over a 7-day treatment period in participants in a stable partnership. Part B assesses the effect of a single dose OXT on sexual arousal, fear and empathy in a clinical setting and is designed for single participants and those in partnerships.

DETAILED DESCRIPTION:
Disruption of the hypothalamic-pituitary axis, caused by inflammation, tumors, or head trauma, can result in arginine vasopressin (AVP) deficiency (AVP-D), formerly known as central diabetes insipidus (cDI). This condition is characterized by polyuria and polydipsia, leading to significant disruptions in the body's fluid balance. Desmopressin, an AVP receptor analogue, is the standard treatment for AVP-D and effectively mitigates these physical symptoms.

However, patients with AVP-D frequently report residual psychological symptoms that remain unaddressed despite desmopressin therapy. These include impaired emotion recognition, reduced empathy, heightened anxiety, social interaction difficulties, and decreased sexual desire-all of which significantly affect their quality of life. Recent data from an international survey of over 1,000 patients with AVP-D reinforce these findings, highlighting the psychosocial burden of this condition.

Oxytocin (OXT), a neuropeptide closely associated with AVP in terms of anatomical location and function, is known to play a critical role in social, emotional, and behavioral regulation. As a "pro-social" hormone, OXT fosters trust, intimacy, attachment, and pair bonding, while also mitigating stress. The proximity of the AVP and OXT systems within the brain suggests that disruptions in one could potentially lead to deficiencies in the other. Supporting this hypothesis, recent research using a novel stimulation test with MDMA demonstrated an OXT deficiency in patients with AVP-D, offering a potential explanation for their observed psychopathology.

OXT's influence extends to sexual well-being, where it has been shown to enhance bonding, intimacy, and the emotional aspects of sexual relationships. Elevated OXT levels are observed during labor, lactation, and sexual arousal, and studies suggest correlations between OXT and orgasm intensity, sexual satisfaction, and partner attachment. While previous studies have examined OXT's effects on social and emotional behavior in healthy individuals, its therapeutic potential in addressing psychological and sexual well-being in AVP-D patients remains unexplored.

This study aims to investigate whether intranasal OXT administration can improve sexual well-being, intimacy, and pair bonding in patients with AVP-D. By addressing an unrecognized OXT deficiency, this research seeks to fill a critical gap in understanding and managing the psychosocial challenges associated with AVP-D.

The trial employs a randomized, double-blind, placebo-controlled, cross-over design and consists of two parts:

1. Part A involves a seven-day treatment with intranasal OXT (24 IU) or placebo in patients with AVP-D and their partners. Participants will self-assess their sexual well-being and intimacy at baseline and after each treatment period, with a three-week washout period between treatments.
2. Part B evaluates the acute effects of a single intranasal OXT dose (24 IU) or placebo on sexual arousal, empathy, fear perception, and hormonal responses to visual stimuli in both single and partnered patients with AVP-D, compared to healthy controls.

This comprehensive approach will provide insights into both the long-term and immediate impacts of OXT therapy, with the ultimate goal of improving quality of life for patients with AVP-D.

ELIGIBILITY:
Inclusion Criteria for healthy controls:

* Adult healthy volunteers aged 18 years and above
* Matched for age, sex, BMI, and menopause/hormonal contraceptives to patients
* No medication, except hormonal contraception
* At least mild impairment in sexual function and satisfaction, defined as an ASEX-score ≥10 points and an NSSS-S score ≤ 48 points
* Only Part A: Participants must be sexually active (at least once a week sexual intercourse) and in a current partnership for at least 6 months

Inclusion criteria for patients:

* Adult patients aged 18 years and above, with a confirmed diagnosis of AVP deficiency based on established criteria
* Stable hormone replacement therapy for at least three months with desmopressin and, in case of additional anterior pituitary deficiencies, with the respective substitution therapies
* At least mild impairment in sexual function and satisfaction, defined as an ASEX-score ≥10 points and an NSSS-S score ≤ 48 points
* Only Part A: Participants must be sexually active (at least once a week sexual intercourse) and in a current partnership for at least 6 months

Exclusion Criteria:

* Pregnancy and breastfeeding within the last eight weeks
* Participation in a trial with investigational drugs within 30 days
* Active substance use disorder within the last six months
* Consumption of alcoholic beverages >15 drinks/week
* Current or previous psychotic disorder (e.g., schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arizona Sexual Experience Scale (ASEX) (Part A) | before treatment and after the 7 day treatement period
  Subjective improvement in sexual well-being and intimacy, defined as a score decrease of 3 or more points on the ASEX (score range: 5-30). Only assessed in Part A
New Sexual Satisfaction Scale (NSSS-S) (Part A) | before treatment and after the 7 day treatement period
  Subjective improvement in sexual well-being and intimacy, with an increase of 3 or more points on the NSSS-S (score range: 12-60). Only assessed in Part A

SECONDARY OUTCOMES:
sexual well-being and intimacy in response to sexual intercourse assesssed by ASEX (Part A) | before treatment and after the 7 day treatement period
  sexual well-being and intimacy in response to sexual intercourse assesssed by ASEX (score range: 5-30, while 30 indicates higher well-being). Comparison of success rates in the primary endpoint between patients with AVP-D and healthy controls
sexual well-being and intimacy in response to sexual intercourse assesssed by NSSS-S (Part A) | before treatment and after the 7 day treatement period
  sexual well-being and intimacy in response to sexual intercourse assesssed by NSSS-S (score range: 12-60, while 60 indicates higher well-being). Comparison of success rates in the primary endpoint between patients with AVP-D and healthy controls
Subjective sexual satisfaction and intimacy of the respective partners (Part A) | before treatment and after the 7 day treatement period
  Levels of sexual satisfaction and intimacy using the short version of the New Sexual Satisfaction Scale (NSSS-S), completed by the partners.
Hormonal response to sexual intercourse (Part B) | at the day of assessement, 2.5 hours
  Area under the salivary cortisol concentration curves in response to sexual Intercourse
Subjective sexual arousal, emotional empathy, fear and fear-induced stress (Part B) | at the day of assessement, 2.5 hours
  Numeric Rating Scales for sexual arousal. Score ranges from 0-75 while 0 indicates minimal sexual arousal
Subjective sexual arousal, emotional empathy, fear and fear-induced stress (PANAS) (Part B) | at the day of assessement, 2.5 hours
  Positive and Negative Affect Schedule (PANAS). Score ranges from 10-50 while higher values represent a greater degree of positive affect.
Subjective sexual arousal, emotional empathy, fear and fear-induced stress (Part B) (SADI) | at the day of assessement, 2.5 hours
  Sexual Arousal and Desire Inventory (SADI); Score ranges from 0-75 while lower scores indicate minimal sexual arousal
Subjective sexual arousal, emotional empathy, fear and fear-induced stress (Part B) (TEQ) | at the day of assessement, 2.5 hours
  Toronto Empathy Questionnaire (TEQ); Score ranges from 0-64 - Higher scores indicate high levels of self-reported empathy while scores below 45 are indicative of below average empathy levels
Subjective sexual arousal, emotional empathy, fear and fear-induced stress (Part B) (STAI-S) | at the day of assessement, 2.5 hours
  State-Anxiety Scale (STAI-S). Total score ranges from 0-40, with higher scores indicating more pronounced anxiety. A score of 20 suggests clinically significant anxiety symptoms.
Autonomic response to sexual arousal and to acute fear-induced stress (Part B) (HR) | during the one day assessment, 2.5 hours
  heart rate measurement
Autonomic response to sexual arousal and to acute fear-induced stress (Part B) (BP) | during the one day assessment, 2.5 hours
  blood pressure measurement
Hormonal response to sexual arousal, emotional empathy and acute fear-induced stress (Part B) | during the one day assessment, 2.5 hours
  Time course of plasma cortisol, oxytocin, neurophysin I, copeptin, prolactin and ACTH levels in response to visual stimuli with erotic, horror and social-positive content
Psychological measures (PFB) | assessed on study inclusion at the baseline visit
  Level of quality of the partnership using the Partnership Questionnaire (PFB). Total score ranges from 0-90; a total score of 54 is considered the threshold for a satisfactory partnership
Psychological measures (SDI-2) | assessed on study inclusion at the baseline visit
  Level of interest in sexual activity using the Sexual Desire Inventory (SDI-2). Total score ranges from 0-78, Dyadic Score : 0-38 & Solitary Score: 0- 40 , higher scores indicating more desire
Psychological measures (SBQ-G) | assessed on study inclusion at the baseline visit
  Level of sexual (dys-)functions using the Sexual Behavior Questionnaire (SBQ-G). Women: 10 items, Men: 11 items; Range: 1-4, with a higher range indicating greater sexual function and desire. Mean Global Index: Sum of 5 items/5 (Median: 2)
Psychological measures (STAI-S) | assessed on study inclusion at the baseline visit
  Level of trait anxiety using the State-Anxiety Scale (STAI-S). 20 items, Total score ranges from 0-40, with higher scores indicating more pronounced anxiety. A score of 20 suggests clinically significant anxiety symptoms.
Psychological measures (TEQ) | assessed on study inclusion at the baseline visit
  Level of emotional empathy using the Toronto Empathy Questionnaire (TEQ). Score ranges from 0-64 while higher scores indicate high levels of self-reported empathy while scores below 45 are indicative of below average empathy levels

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. MD, Principal Investigator — Universitätsspital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland